CLINICAL TRIAL: NCT05911035
Title: Post COVID-19 Acute Mucormycosis in Critical Care Settings in Egypt: A Single-Center Experience
Brief Title: Post-COVID-19 Mucormycosis in Critical Care
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ayman Magd Eldin Mohammad Sadek, Associate Professor of Internal Medicine, Zagazig University
Other Study IDs: ZU-IRB#9491/26-4-2022
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Mucormycosis; Rhinocerebral (Etiology); Post COVID-19 Condition, Unspecified
Keywords: Mucormycosis; Post COVID-19; Cutaneous infection; Ocular infection; Sinus infection
MeSH Terms: conditions — Mucormycosis; Eye Infections; Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Mucormycosis is a life-threatening opportunistic fungal infection. Despite mucormycosis having existed for decades, it has gained notice of its widespread in many parts of the world during the second wave of the coronavirus disease 2019 (COVID-19) pandemic. The study aimed to determine the in-hospital outcomes of post-COVID-19 mucormycosis during the intensive care unit (ICU) stay in Egypt.

Methods: This prospective cohort study included all patients admitted to the Medical ICU of the University Hospital who developed Mucormycosis with a history of previous COVID-19 infection. Clearance of previous COVID-19 was confirmed using PCR and high-resolution computed tomography (CT) on the chest before admission.

DETAILED DESCRIPTION:
Study design, settings, and participants This prospective cohort study was conducted in the medical ICU of the Zagazig University Hospital, Egypt, comprising 150 Post COVID-19 patients who developed Mucormycosis infection.

The investigators take the approval of the Institutional Review Board (IRB) ethical committee under code (ZU-IRB#9491/26-4-2022). The study was conducted under the guidance of the Declaration of Helsinki. Written informed consent was taken from all patients or first-degree relatives in case of altered sensorium.

The inclusion criteria were all patients aged 18 or older, of both genders, and confirmed previous COVID-19 with Mucormycosis infection were included in this study. We excluded patients with other fungal infections post-COVID-19 or Mucormycosis infection without previous COVID-19.

Process For all cases, the first step was to perform a polymerase chain reaction (PCR) to exclude current COVID-19 on admission and high-resolution computed tomography (CT) on the chest.

The complete medical history was also recorded of all patients, including demographic details (age, gender, residence, and smoking) and the risk factors, such as diabetes mellitus (DM), hypertension, chronic kidney disease (CKD), and other comorbidities).

Routine laboratory investigations were conducted, including complete blood count (CBC), liver functions, kidney functions, C-reactive protein (CRP), and arterial blood gases (ABG) daily. Also, Glycated hemoglobin (HbA1c), D-Dimer, Procalcitonin (PCT), Ferritin at admission, sodium (Na), and potassium (K) every four hours. In addition to specific laboratory investigations like a cluster of differentiation (CD4/CD8) ratio on admission and interleukin 6 (IL6) on admission and after three days. The patient also had further investigations, such as electrocardiography (ECG).

Regarding imaging, routine studies like abdominal ultrasonography (US) and echocardiography or specific for mucormycosis like CT or magnetic resonance imaging (MRI) for brain and nasal sinuses were conducted. For patients who needed surgical debridement, preoperative viral markers (HCV antibody, HBs antigen, HIV antibody) were drawn, and intraoperative biopsies were taken for histopathological examination. Patients initially received conventional Amphotericin B, while in case of therapy complications, the treatment is converted to liposomal Amphotericin B.

ELIGIBILITY:
Inclusion Criteria:

* confirmed previous COVID-19 infection with new mucormycosis infection

Exclusion Criteria:

* other fungal infections post-COVID-19 or mucormycosis infections without previous COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a history of previously cleared COVID-19 infection who were admitted to critical care with newly developed mucormycosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 48 weeks
  mortality rate of patients with mucormycosis in the critical care

SECONDARY OUTCOMES:
Complications | 48weeks
  complications arise from the treatment with Amphotericin B

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sadek, MD, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Human Medicine, Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No